CLINICAL TRIAL: NCT02350231
Title: Progesterone Vaginal Pessary for Prevention of Preterm Twin Birth
Acronym: PPPTP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Sohag University (Other)
Responsible Party: Principal Investigator, Omar Mamdouh Shaaban, Professor of Obstetrics and Gynecology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Progesterone vaginal pessary
Record Dates: First submitted 2015-01-05; First posted 2015-01-29 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Preterm Birth
Keywords: preterm birth; Twin pregnancy; progesterone
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The progesterone vaginal pessary group (Active Comparator): Where they will have progesterone vaginal pessary (Prontogest 400 mg) daily at bed time from 28 weeks of pregnancy till delivery in addition to tonic and calcium
  Interventions: Drug: The progesterone vaginal pessary
- Tonics group (Placebo Comparator): Where they will receive only tonics and calcium from 28 weeks of pregnancy till delivery
  Interventions: Drug: Tonics group

INTERVENTIONS:
Drug: The progesterone vaginal pessary — Those patients will receive progesterone vaginal pessary for prevention of preterm delivery in twins pregnancy
  Other Names: Active drug treatment
  Arms: The progesterone vaginal pessary group
Drug: Tonics group — Those patients will receive only tonics
  Other Names: Placepo
  Arms: Tonics group

SUMMARY:
Multiple pregnancies accounted for 1 - 6 % of all births in UK during 2007. More than 98% of these multiple births being twin births . Preterm birth defined as birth occurring prior to 37 weeks of gestation and it was about 15 % of pregnancies in developed world and 12.7 % in the United States.

Preterm birth is the leading cause of infant and neonatal mortality. Premature neonates are at increased risk of developing respiratory distress syndrome, sepsis, intraventricular hemorrhage, and necrotizing enterocolitis.

Twin pregnancy is considered one of the important risk factors of preterm birth. Over distension of uterus may be one of the etiological factors for preterm birth. However, no definite effective interventions have been shown to prevent preterm delivery in twin pregnancy.

Three large randomized trials suggested that progesterone might prevent preterm delivery in high-risk singleton pregnancy especially those with previous preterm delivery or short cervix might be reduced by antenatal progesterone.

Fonseca et al (2007) concluded that women with short cervix are less likely to deliver preterm ≤34 weeks if they are treated with vaginal progesterone.

ELIGIBILITY:
Inclusion Criteria:

1. Diamniotic twin pregnancy
2. Gestational age ± 28 weeks.

Exclusion Criteria:

1. Higher multiple pregnancy
2. IUFD of one or both fetuses
3. Any congenital anomalies
4. IUGR or discordant twins
5. PROM
6. If there is any contraindication to progesterone treatment
7. Women who did performed cervical cerclage in the current pregnancy
8. Difficult in follow up for the pregnant women as (living faraway area, or difficult transportion, etc).
9. Threatened preterm labor.
10. Polyhydromnis.
11. Other medical disorder with pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Time of delivery | from 28 weeks till delivery

SECONDARY OUTCOMES:
Mode of delivery | from 28 weeks till delivery
Birth weight | at time of delivery
The need for neonatal intensive care incubator. | after delivery